CLINICAL TRIAL: NCT02997800
Title: The Effect of Intraoperative Labetalol on Time to Discharge and Hemodynamic Stability in Laparoscopic Cholecystectomy
Brief Title: The Effect of Intraoperative Labetalol on Time to Discharge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Robert Tanzola (Other)
Responsible Party: Sponsor-Investigator, Dr. Robert Tanzola, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANAE-219-12
Record Dates: First submitted 2016-12-08; First posted 2016-12-20 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Bloodpressure; Heart Rate
MeSH Terms: interventions — esmolol; Labetalol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Esmolol (Experimental): Esmolol infusion and 1 ml saline infusion
  Interventions: Drug: Esmolol; Other: 1 ml saline infusion
- Labetalol (Experimental): Labetalol Bolus and saline infusion
  Interventions: Drug: Labetalol; Other: saline infusion
- Fentanyl (Active Comparator): Fentanyl Bolus and saline infusion
  Interventions: Drug: Fentanyl; Other: saline infusion

INTERVENTIONS:
Drug: Esmolol — Following induction and intubation, any increase in heart rate (HR) or mean arterial pressure (MAP) >20% of baseline will be treated with an initial intravenous bolus of esmolol 30 mg IV (30 mg in 5 ml of normal saline). An intravenous esmolol infusion will be initiated at 5mcg/kg/min after the first intravenous bolus dose and will be titrated up by 5mcg/kg/min each time HR or MAP >20% of baseline. An intravenous bolus of placebo (normal saline 1 ml) will be administered whenever a change to the infusion rate is made.
  Arms: Esmolol
Drug: Labetalol — Following induction and intubation, any increase in heart rate (HR) or mean arterial pressure (MAP) >20% of baseline will be treated with an initial intravenous bolus of labetalol 10 mg IV (10 mg in 5 ml of normal saline). Any further increases in HR or MAP >20% of baseline will be treated with intravenous boluses of labetalol 5 mg in 1 ml every 5 minutes as needed. An intravenous placebo infusion (normal saline) will be initiated at 5 mcg/kg/min after the first intravenous bolus dose and will be titrated up by 5 mcg/kg/min each time an additional intravenous bolus is given.
  Arms: Labetalol
Drug: Fentanyl — Following induction and intubation, any increase in heart rate (HR) or mean arterial pressure (MAP) >20% of baseline will be treated with an initial intravenous bolus of fentanyl 50 mcg IV (50 mcg in 5 ml of normal saline). Any further increases in HR or MAP >20% of baseline will be treated with intravenous boluses of fentanyl 25 mcg in 1 ml every 5 minutes as needed. An intravenous placebo infusion (normal saline) will be initiated at 5 mcg/kg/min after the first intravenous bolus dose and will be titrated up by 5 mcg/kg/min each time an additional intravenous bolus is given.
  Arms: Fentanyl
Other: saline infusion — An intravenous placebo infusion (normal saline) will be initiated at 5 mcg/kg/min after the first intravenous bolus drug dose (fentanyl or labetalol depending upon randomization) and will be titrated up by 5 mcg/kg/min each time an additional intravenous bolus is given.
  Arms: Fentanyl; Labetalol
Other: 1 ml saline infusion — Every time the infusion rate of esmolol is changed, 1 ml of normal saline will be infused.
  Arms: Esmolol

SUMMARY:
Patients coming for surgery often receive opioid medications, like fentanyl, to treat pain. Opioids however have many unpleasant side effects including nausea and vomiting, itching, sedation, and decreased breathing. During laparoscopic surgery increases in heart and blood pressure are often attributed to pain. It has been shown that by treating these changes with medications such as esmolol, instead of opioids, side effects and time to discharge from hospital can be reduced. Labetalol is a drug that is similar to esmolol but may have advantages over it. It is more effective at controlling both heart rate and blood pressure and it is easier and less costly to use. This study is investigating labetalol in patients having laparoscopic gallbladder surgery and comparing it to esmolol and fentanyl. Patients will be treated with one of these drugs during surgery to control heart rate and blood pressure and the effects on time to discharge, pain scores, frequency of side effects, and narcotic requirements will be observed in the recovery room. It is thought that labetalol will be shown to be as effective as esmolol and that both drugs that minimize fentanyl will show reduced time to discharge, fewer side effects, and effective treatment of heart rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo elective ambulatory laparoscopic cholecystectomy under general anesthesia
* American Society of Anesthesiologist's Status ASA) 1-3
* able to understand and sign informed consent

Exclusion Criteria:

* known allergy to any of the study medications including beta blockers, fentanyl, acetaminophen, non-steroidal anti-inflammatories or local anesthetics
* chronic use of beta-adrenergic receptor antagonists or opioids
* conversion to open cholecystectomy
* History of renal, hepatic or cardiac failure, reactive airway disease
* Medical history that in the investigator's judgement would interfere with the protocol or assessments
* Unable to understand pain assessment
* Failure to give informed consent
* pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-11; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Length of stay in the post-anesthesia care unit (PACU) | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  time from arrival in PACU after surgery until discharge from PACU

SECONDARY OUTCOMES:
Intraoperative Heart Rate (HR) | intraoperatively-from anesthesia induction to the surgery completion (wound closure) -approximately 45 min.
  heart rate (beats per min.)
Intraoperative mean arterial pressure (MAP) | intraoperatively-from anesthesia induction to the surgery completion (wound closure)-approximately 45 min.
  blood pressure (mmHg)
postoperative nausea and vomiting (PONV) in PACU | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  incidence of nausea and vomiting
pain scores | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  pain scores visual analogue scale (VAS)
fentanyl required | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  total fentanyl required mcg
adverse effects | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  Any reported adverse effects or complications
postoperative heart rate | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  heart rate (beats per min)
postoperative mean arterial pressure (MAP) | The time-frame between entry to PACU and discharge from PACU (approximately 1.5 hours).
  blood pressure (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tanzola, MD, FRCPC, Principal Investigator — Queen's University-Anesthesiology
Locations (1):
- Queen's University, Department of Anesthesiology, Kingston, Ontario, Canada